CLINICAL TRIAL: NCT00191464
Title: Long-Term Effects of Insulin Plus Metformin Regimens on the Overall and Postprandial Glycemic Control of Patients With Type 2 Diabetes: A Comparison of Premeal Insulin Lispro Mixtures to Once-Daily Insulin Glargine
Brief Title: Long-Term Effects of Insulin Plus Metformin Regimens on the Overall and Postprandial Glycemic Control of Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6146; F3Z-MC-IOOI
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Metformin

INTERVENTIONS:
Drug: premeal insulin lispro mixtures
Drug: insulin glargine
Drug: metformin

SUMMARY:
The primary objective of this study is to show that a prandial insulin regimen, consisting of premeal insulin lispro "mid mixture" (or a combined regimen of insulin lispro "mid mixture" and insulin lispro "low mixture") plus metformin will result in significantly better overall glycemic control (lower HbA1c) at endpoint than once-daily insulin glargine plus metformin. Insulin lispro "mid mixture" consists of 50% insulin lispro and 50% NPL. Insulin lispro "low mixture" consists of 25% insulin lispro and 75% NPL.

In a substudy of approximately 60 patients, additional data will be collected on markers associated with risk of atherosclerosis or cardiovascular disease in the context of a controlled, outpatient, high-fat test meal.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes (World Health Organization [WHO] classification
* Have used one or more of the following oral anti-hyperglycemic medications-metformin or second-generation sulfonylurea (for example, glibenclamide, glyburide, glipizide, gliclazide, glimepiride) alone or in combination with one or two insulin injections per day for at least 3 months immediately prior to entering the study. Patients using more than 2 insulin injections per day or subcutaneous insulin infusion prior to the study will not be eligible to participate.
* Have a hemoglobin A1c between 6.5% and 11%, inclusive, according to the central laboratory at Visit 1.
* Have clinically acceptable LDL-C, in the investigator's opinion, at Visit 1.
* As determined by the investigator, are capable and willing to learn how to use the insulin injection pens; comply with their prescribed diet, exercise, and medication regimen; perform self-monitoring of blood glucose; and use the patient diary as required for this protocol.

Exclusion Criteria:

* Have hypersensitivity to metformin or a known allergy to metformin hydrochloride, insulin lispro MM, insulin lispro LM, or insulin glargine, or excipients contained in these products.
* Have known metabolic or lactic acidosis.
* Have a history of renal transplantation or are currently receiving renal dialysis or have serum creatinine greater than or equal to 135 micromol/L (1.5 mg/dL) for males and greater than or equal to 110 micromol/L (1.2 mg/dL) for females.
* Have cardiac disease with functional status that is Class III or IV
* Have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, or alanine transaminase (ALT) greater than three times the upper limit of the reference range as defined by the central laboratory.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320
Dates: Start 2003-12; Study Completion 2005-09

PRIMARY OUTCOMES:
HbA1C

SECONDARY OUTCOMES:
General inflammation (hsCRP)
High-density lipoprotein cholesterol
Total cholesterol
Triglycerides
Estimates of low-density lipoprotein cholesterol
Nuclear magnetic resonance [NMR] analysis of lipids
Oxidized LDL
Lipoproteins and apoproteins
Fibrinogen
Blood glucose levels (based on self-monitoring)
Insulin dose
Weight
Frequency and incidence of hypoglycemia
Safety
General well-being
Pilot two questionnaires for microvascular complications
Coagulopathy factors [substudy]
Surrogate measure of vascular reactivity [substudy]
Inflammatory markers [substudy]
Production of advanced glycation end-products [substudy]
Generation of oxidative species [substudy]
Lipids in various fractions [substudy]
Retinyl ester measurements in various fractions [substudy]
Composition of triglyceride-rich lipoproteins [substudy]
Compartmental modeling of postprandial lipemia [substudy]
Apolipoproteins [substudy]

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lebanon, New Hampshire, United States
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Leonards, New South Wales, Australia
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki, Greece
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mumbai, Maharstra, India
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Den Helder, Netherlands
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oleśnica, Poland
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ponce, Puerto Rico

REFERENCES:
- [Background] Robbins DC, Beisswenger PJ, Ceriello A, Goldberg RB, Moses RG, Pagkalos EM, Milicevic Z, Jones CA, Sarwat S, Tan MH. Mealtime 50/50 basal + prandial insulin analogue mixture with a basal insulin analogue, both plus metformin, in the achievement of target HbA1c and pre- and postprandial blood glucose levels in patients with type 2 diabetes: a multinational, 24-week, randomized, open-label, parallel-group comparison. Clin Ther. 2007 Nov;29(11):2349-64. doi: 10.1016/j.clinthera.2007.11.016. PMID 18158076
- [Result] Hirsch IB, Yuan H, Campaigne BN, Tan MH. Impact of prandial plus basal vs basal insulin on glycemic variability in type 2 diabetic patients. Endocr Pract. 2009 May-Jun;15(4):343-8. doi: 10.4158/EP08308.ORR. PMID 19454394
- [Result] Chan JY, Leyk M, Frier BM, Tan MH. Relationship between HbA1c and hypoglycaemia in patients with type 2 diabetes treated with different insulin regimens in combination with metformin. Diabetes Metab Res Rev. 2009 Mar;25(3):224-31. doi: 10.1002/dmrr.929. PMID 19156705
- [Result] Shrom D, Sarwat S, Ilag L, Bloomgarden ZT. Does A1c consistently reflect mean plasma glucose? J Diabetes. 2010 Jun;2(2):92-6. doi: 10.1111/j.1753-0407.2010.00066.x. Epub 2010 Jan 22. PMID 20923490
- [Result] Sarwat S, Ilag LL, Carey MA, Shrom DS, Heine RJ. The relationship between self-monitored blood glucose values and glycated haemoglobin in insulin-treated patients with Type 2 diabetes. Diabet Med. 2010 May;27(5):589-92. doi: 10.1111/j.1464-5491.2010.02955.x. PMID 20536957
- [Derived] Beisswenger PJ, Brown WV, Ceriello A, Le NA, Goldberg RB, Cooke JP, Robbins DC, Sarwat S, Yuan H, Jones CA, Tan MH; IOOI Study Investigators. Meal-induced increases in C-reactive protein, interleukin-6 and tumour necrosis factor alpha are attenuated by prandial + basal insulin in patients with Type 2 diabetes. Diabet Med. 2011 Sep;28(9):1088-95. doi: 10.1111/j.1464-5491.2011.03324.x. PMID 21517955